CLINICAL TRIAL: NCT00836914
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Two-Period Crossover Study to Investigate the Safety of CAL-101 in Allergic Rhinitis Subjects and Effects on the Response to Environmental Chamber Allergen Challenge
Brief Title: Study to Investigate Effects of CAL-101 in Subjects With Allergic Rhinitis Exposed to Allergen in an Environmental Chamber
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 101-04
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2013-01

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis; Allergy; Phosphatidylinositol 3-kinase
MeSH Terms: conditions — Rhinitis, Allergic; Hypersensitivity | interventions — idelalisib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAL-101 (Active Comparator)
  Interventions: Drug: CAL-101
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CAL-101 — CAL-101 100mg capsules administered orally twice a day (BID) for 7 days
  Other Names: Idelalisib; GS-1101
  Arms: CAL-101
Drug: Placebo — Placebo capsules administered orally BID for 7 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and effect of CAL-101 in subjects with allergic rhinitis.

DETAILED DESCRIPTION:
A Phase I, randomized, double-blind crossover study of CAL-101, an oral inhibitor of phosphatidylinositol 3-kinase (PI3K) delta, in patients with allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

1. Age > or = 18 and < or = 55 years
2. Has a history of seasonal allergic rhinitis for at least 2 years
3. Has sensitivity to grass pollen demonstrated by a positive response to skin prick testing
4. Has a positive Radio Allergen Sorbent Test (> or = class 2) for grass pollen during the previous 12 months or at screening
5. Is otherwise healthy, that is, free from clinically significant illness or disease as determined by medical history, physical examination and laboratory tests, including a normal 12-lead electrocardiogram (ECG)
6. Has no conditions which would make the subject unlikely to be able to remain in the allergen challenge chamber for 4 hours
7. Is available to complete all study procedures
8. Is able to provide written informed consent, including compliance with the requirements and restrictions listed in the consent form

Exclusion Criteria:

1. Is a female of childbearing potential (non-childbearing potential means documented surgery resulting in infertility or postmenopausal with no menses for at least 1 year)
2. History of chronic nasal or upper respiratory tract symptoms or disorders other than allergic rhinitis
3. History of nonallergic rhinitis, chronic sinusitis or severe asthma
4. Has a nasal condition likely to affect the outcome of the study, i.e. nasal septal perforations, nasal polyps, sinus disease, chronic nasal obstruction, or other nasal diseases
5. Is currently taking regular medication, whether prescribed or not, including corticosteroids, vitamins, macrolides, anti-fungal agents and herbal remedies, e.g. St. John's Wort. Paracetamol (< or = 2g/day) and as needed use of short-acting B2-agonists are allowed.
6. Has taken a prohibited medication within the specified interval prior to Visit 1:

   * Corticosteroids (depot, 90 days; systemic, 30 days; dermatologic 14 days)
   * Chromones (14 days)
   * Antihistamines (nasal and long-acting oral, 10 days; shorting-acting oral, 2 days; ocular, 3 days)
   * Decongestants (3 days)
   * Leukotriene modifiers (10 days)
   * Anticholinergics (7 days)
   * Opthalmic nonsteroidal
   * anti-inflammatory drugs (3 days)
   * Nasal-ophthalmic wash solutions (12 hr)
   * Immunotherapy (12 hr)
7. Is currently being treated with a medication that induces or inhibits cytochrome P450 (CYP)3A

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2009-02; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety CAL-101 using adverse events, vital signs, clinical laboratory tests, spirometry and ECG | Baseline to Day 35

SECONDARY OUTCOMES:
Change from baseline in total nasal symptom score | Baseline to Day 35

CONTACTS AND LOCATIONS:
Overall Officials: Friedrich Horak, MD, Principal Investigator — Vienna Challenge Chamber
Locations (1):
- Vienna Challenge Chamber, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Derived] Horak F, Puri KD, Steiner BH, Holes L, Xing G, Zieglmayer P, Zieglmayer R, Lemell P, Yu A. Randomized phase 1 study of the phosphatidylinositol 3-kinase delta inhibitor idelalisib in patients with allergic rhinitis. J Allergy Clin Immunol. 2016 Jun;137(6):1733-1741. doi: 10.1016/j.jaci.2015.12.1313. Epub 2016 Feb 23. PMID 26915677